CLINICAL TRIAL: NCT03422406
Title: A Prospective Observational Study on Health Effect of Excessive Iodine Exposure in Pregnancy
Brief Title: Research on Excessive Iodine Status in Pregnancy
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Liuyanping
Record Dates: First submitted 2018-01-24; First posted 2018-02-05 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Excessive Iodine Status; Thyroid Dysfunction, Antepartum; Pregnancy Related; Neonatal Disorder
Keywords: Iodine excess; Cause; Pregnancy; Urinary iodine concentration; Serum iodine concentration; Breast milk iodine concentration
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine for urinary iodine concentration analysis;serum for serum iodine concentration analysis; maternal breast milk for colostrum iodine concentration analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HH group: Group (participants) with pre-gestational history of undergoing hysterosalpingography (HSG) using an oil-soluble iodinated contrast medium
  Interventions: Other: Dietary iodine intake restriction
- Non-HH group: Group (participants) without pre-gestational history of undergoing hysterosalpingography (HSG)
  Interventions: Other: Dietary iodine intake restriction

INTERVENTIONS:
Other: Dietary iodine intake restriction — All subjects with excessive iodine load were recommended by nutritionists to restrict dietary iodine intake, and resume iodine-containing supplements and foods until their iodine status return to normal. However, in this observational study, the intervention was a regular management in prenatal care, and not assigned by investigator of the study.

SUMMARY:
To explore main cause and health impact of iodine excess during pregnancy, we performed iodine evaluation for 390 consecutive pregnant women from January 1st, 2016 to December 31st, 2016. Among them, 18 women (4.62%) with apparently elevated urinary iodine concentration (UIC) were enrolled onto this study for subsequent follow-up. History of high iodine exposure was collected from all participants. Parameters about iodine status were monitors until termination of pregnancy, and dietary iodine intake condition and thyroid function were also evaluated.

DETAILED DESCRIPTION:
A prospective follow-up was arranged for the 18 pregnant women with excessive iodine status. History of iodine exposure (including hysterosalpingography (HSG) using an oil-soluble iodinated contrast medium, examination by computed tomography scan with contrast, administration of amiodarone, history of receiving radioiodine therapy, etc.) was collected from all participants. Evaluation of dietary iodine intake was performed through a 72-hour dietary recall.The serum iodine concentration (SIC) and urinary iodine concentration (UIC) were monitored continuously in the whole course of pregnancy. All subjects with excessive iodine load were recommended by nutritionists to have their dietary iodine intake restricted, and resume iodine-containing supplements and foods until the UIC<250 μg/L and SIC≤90 μg/L. After delivery, maternal colostrum iodine concentration and neonatal iodine status (including neonatal UIC, condition of congenital hypothyroidism screening tests, and thyroid physical examination) were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with apparently elevated urinary iodine concentration (UIC ≥250μg/L) and serum iodine concentration (SIC>90μg/L) were enrolled in this study.

Exclusion Criteria:

* Subject who did not sign the informed consent or whose clinical date was not intact was excluded in our study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All enrolled pregnant women will be from urban area of Beijing, whose dietary iodine intake and pre-gestational history of iodine exposure will be reviewd in detail.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
prevalence of adverse pregnancy outcome | 6-9 months post identification of maternal iodine excess
  prevalence of stillbirth, abortion and other adverse pregnancy outcome
composite neonatal outcome | 6-9 months post identification of maternal iodine excess
  Apgar scores, birth weight of the neonates,and prevalence of thyroid dysfunction in neonates

SECONDARY OUTCOMES:
prevalence of maternal thyroid dysfunction in pregnancy | through study completion, about 6-9 months post identification of maternal iodine excess
  Laboratory reference ranges of TSH during pregnancy were 0.1~2.5 mIU/L for the first trimester, 0.2~3.0 mIU/L for the second trimester and 0.3~3.0 mIU/L for the third trimester.Prevalence of TSH elevation during pregnancy will be summarized.
prevalence of neonatal iodine excess | within 1 week after birth
  urinary iodine concentration will be examined for all neonates born to women with iodine excess in pregnancy, and prevalence of neonatal urinary iodine concentration ≥ 200μg/L will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zhang, MD, Study Chair — Department of academic research,Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sun D, Codling K, Chang S, Zhang S, Shen H, Su X, Chen Z, Scherpbier RW, Yan J. Eliminating Iodine Deficiency in China: Achievements, Challenges and Global Implications. Nutrients. 2017 Apr 5;9(4):361. doi: 10.3390/nu9040361. PMID 28379180
- [Result] Alexander EK, Pearce EN, Brent GA, Brown RS, Chen H, Dosiou C, Grobman WA, Laurberg P, Lazarus JH, Mandel SJ, Peeters RP, Sullivan S. 2017 Guidelines of the American Thyroid Association for the Diagnosis and Management of Thyroid Disease During Pregnancy and the Postpartum. Thyroid. 2017 Mar;27(3):315-389. doi: 10.1089/thy.2016.0457. PMID 28056690
- [Result] Xiao Y, Sun H, Li C, Li Y, Peng S, Fan C, Teng W, Shan Z. Effect of Iodine Nutrition on Pregnancy Outcomes in an Iodine-Sufficient Area in China. Biol Trace Elem Res. 2018 Apr;182(2):231-237. doi: 10.1007/s12011-017-1101-4. Epub 2017 Aug 2. PMID 28770411
- [Result] So S, Yamaguchi W, Tajima H, Nakayama T, Tamura N, Kanayama N, Tawara F. The effect of oil and water-soluble contrast medium in hysterosalpingography on thyroid function. Gynecol Endocrinol. 2017 Sep;33(9):682-685. doi: 10.1080/09513590.2017.1307960. Epub 2017 Apr 17. PMID 28412871
- [Result] Kaneshige T, Arata N, Harada S, Ohashi T, Sato S, Umehara N, Saito T, Saito H, Murashima A, Sago H. Changes in serum iodine concentration, urinary iodine excretion and thyroid function after hysterosalpingography using an oil-soluble iodinated contrast medium (lipiodol). J Clin Endocrinol Metab. 2015 Mar;100(3):E469-72. doi: 10.1210/jc.2014-2731. Epub 2014 Dec 29. PMID 25546154
- [Result] Satoh M, Aso K, Katagiri Y. Thyroid Dysfunction in Neonates Born to Mothers Who Have Undergone Hysterosalpingography Involving an Oil-Soluble Iodinated Contrast Medium. Horm Res Paediatr. 2015;84(6):370-5. doi: 10.1159/000439381. Epub 2015 Sep 25. PMID 26402613
- [Result] Mekaru K, Kamiyama S, Masamoto H, Sakumoto K, Aoki Y. Thyroid function after hysterosalpingography using an oil-soluble iodinated contrast medium. Gynecol Endocrinol. 2008 Sep;24(9):498-501. doi: 10.1080/09513590802246364. PMID 18958768
- [Result] Omoto A, Kurimoto C, Minagawa M, Shozu M. A case of fetal goiter that resolved spontaneously after birth. J Clin Endocrinol Metab. 2013 Oct;98(10):3910-1. doi: 10.1210/jc.2013-1066. Epub 2013 Aug 26. No abstract available. PMID 23979952